CLINICAL TRIAL: NCT05134584
Title: Efficacy and Safety of Linaclotide in Patients With Overlap of Functional Dyspepsia and Constipation-predominant Irritable Bowel Syndrome
Brief Title: Efficacy of Linaclotide in Patients With Overlapping Functional Gastrointestinal Disorders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, professor,chief physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RenJiH211012
Record Dates: First submitted 2021-11-14; First posted 2021-11-26 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Functional Dyspepsia; Constipation-predominant Irritable Bowel Syndrome
Keywords: functional dyspepsia; irritable bowel syndrome; constipation; linaclotide; lactulose
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation | interventions — linaclotide; Lactulose; Omeprazole; itopride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and investigators were not masked to group assignment. An independent statistician was masked for the data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- linaclotide (Experimental): Patients in linaclotide group were given with oral, once daily 290 μg linaclotide for consecutively 4 weeks, along with once daily 20 mg omeprazole, three times daily 50 mg Itopride, for the first ten days of the treatment.
  Interventions: Drug: Linaclotide; Drug: Omeprazol; Drug: Itopride
- lactulose (Active Comparator): Patients in Lactulose group were given with oral, once daily 20 mL Lactulose for 4 weeks, along with once daily 20 mg omeprazole, three times daily 50 mg Itopride, for the first ten days of the treatment.
  Interventions: Drug: Lactulose; Drug: Omeprazol; Drug: Itopride

INTERVENTIONS:
Drug: Linaclotide — 290μg once daily, 4 weeks
  Other Names: Linzess
  Arms: linaclotide
Drug: Lactulose — 20mL once daily, 4 weeks
  Other Names: Duphalac
  Arms: lactulose
Drug: Omeprazol — 20mg twice daily for the first 10 days
Drug: Itopride — 50mg three times daily for the first 10 days

SUMMARY:
This study aims to assess the efficacy and safety of linaclotide in patients with overlapping symptoms of both functional dyspepsia (FD) and constipation-predominant irritable bowel syndrome (IBS-C).

DETAILED DESCRIPTION:
After being informed about the content and risks of the research, all eligible patients giving written informed consent will be randomly allocated in a 2:1 ratio to linaclotide (290μg, once daily) or lactulose (20mL, once daily). Treatment will last consecutively for 4 weeks, and patients' symptoms will be assessed before and after four-week treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients
2. Diagnosis of FD (including postprandial distress syndrome [PDS] with or without epigastric pain syndrome [EPS]) (Rome Ⅲ criteria)
3. Diagnosis of IBS-C (Rome Ⅲ criteria)

Exclusion Criteria:

1. Helicobacter Pylori infection
2. GI symptoms caused by taking non-steroidal anti-inflammatory drugs or other agents
3. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Treatment satisfaction assessed by the VAS | Week 4
  Treatment satisfaction will be assessed by the Visual Analogue Scale: score 0=not at all, 1=partial relief of general GI symptoms, 2=complete relief of general GI symptoms.

SECONDARY OUTCOMES:
Changes in stool frequency | Baseline and Week 4
  Stool frequency will be assessed using bowel movement (BM), spontaneous bowel movement (SBM), complete spontaneous bowel movement (CSBM) during the past 7 days.
  Change = (Week 4 Score - Baseline Score).
Changes in stool consistency | Baseline and Week 4
  Stool consistency will be assessed using Bristol Stool Form Scale (BSFS), which contains 7 types of stool consistency.
  Change = (Week 4 Score - Baseline Score).
Changes in defecation straining score | Baseline and Week 4
  Defecation straining score will be assessed using six-point scale (score 0 = effortless, 5 = extremely laborious).
  Change = (Week 4 Score - Baseline Score).
Changes in defecation time | Baseline and Week 4
  Defecation time will be assessed using approximate duration: less than 15 minutes, 15-30 minutes, more than 30 minutes.
Changes in sensation of complete evacuation | Baseline and Week 4
  Sensation of complete evacuation will be assessed using five-point scale (score 0 = not at all, 4 = complete totally).
  Change = (Week 4 Score - Baseline Score).
Changes in lower abdominal discomfort | Baseline and Week 4
  Lower abdominal discomfort will be assessed using six-point scale (score 0 = not at all, 5 = extremely severe).
  Change = (Week 4 Score - Baseline Score).
Changes in lower abdominal pain | Baseline and Week 4
  Lower abdominal pain will be assessed using six-point scale (score 0 = not at all, 5 = extremely severe).
  Change = (Week 4 Score - Baseline Score).
Changes in FD symptoms | Baseline and Week 4
  FD symptoms will be assessed using Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM).
  Change = (Week 4 Score - Baseline Score).
Changes in the anxiety status | Baseline and Week 4
  The anxiety status will be assessed using the Generalized Anxiety Disorder scale (GAD-7).
  Change = (Week 4 Score - Baseline Score).
Changes in the depression status | Baseline and Week 4
  The depression status will be assessed using the Patient Health Questionnaire (PHD-9).
  Change = (Week 4 Score - Baseline Score).

CONTACTS AND LOCATIONS:
Overall Officials: Shengliang Chen, Principal Investigator — RenJi Hospital
Locations (1):
- RenJiH, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Cheng L, Wang Q, Wu B, Yan X, Xu P, Qiu H, Chen S. Efficacy of Linaclotide in Functional Dyspepsia and Constipation-Predominant Irritable Bowel Syndrome Overlap: A Randomized Trial. J Gastroenterol Hepatol. 2025 May;40(5):1119-1127. doi: 10.1111/jgh.16925. Epub 2025 Mar 13. PMID 40079184